CLINICAL TRIAL: NCT00267566
Title: Strongest Families (Formerly Family Help Program): Primary Care Delivery by Telephone for Psychological and Behavioural Problems (Pediatric Anxiety)
Brief Title: Strongest Families (Formerly Family Help Program): Pediatric Anxiety
Acronym: FHP-ANX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2234a; CIHR CAHR-43273
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): 50% random assignment to receive Family Help Anxiety Treatment
  Interventions: Behavioral: Strongest Families (formerly Family Help Program): Anxiety Program
- Control (Experimental): 50% random assignment to control group to receive usual/standard care for anxiety
  Interventions: Behavioral: Strongest Families (formerly Family Help Program): Anxiety Program

INTERVENTIONS:
Behavioral: Strongest Families (formerly Family Help Program): Anxiety Program — Evidence-based psychological and behavioural distance intervention
  Other Names: Strongest Families (formerly Family Help Program)

SUMMARY:
The purpose of the Strongest Families (formerly Family Help Program)is to evaluate the effectiveness of the Strongest Families distance intervention compared to usual or standard care that is typically provided to children with mild to moderate Anxiety symptomology. This is a single-center trial based at the IWK Health Center. The primary outcome is change in diagnosis.

DETAILED DESCRIPTION:
The purpose of the Strongest Families (formerly Family Help Program)is to deliver, primary care mental health services to children and their families in the comfort and privacy of their own home. Approximately 128 children (6-12 years of age)suffering from mild to moderate (but clinically significant) symptoms of pediatric anxiety will be randomized.

The intervention is delivered from a distance, using educational materials (manuals, video-tapes, audio-tapes) and telephone consultation with a trained paraprofessional "coach" who is supervised by a licensed health care professional. The telephone coach delivers consistent care based on written protocols, with on-going evaluation by a professional team.

Fifty percent of the eligible participants will receive Strongest Families (formerly Family Help Program) telephone-based treatment and 50% will be referred back to their family physician to receive standard care as determined by that physician. Those receiving standard care will be evaluated for outcome results and then compared to the Family Help treated participants. It is anticipated that Family Help treatment will be proven to be as or more effective than standard care.

ELIGIBILITY:
Inclusion Criteria:

* child 6 to 12 years of age
* child had Anxiety symptoms for 6 months or longer
* access to a telephone in the home
* speak and write english
* mild to moderate anxiety symptomology

Exclusion Criteria:

* severe anxiety symptomology
* received similar intervention within past 6 months
* excessive anxiety following a significant traumatic event

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2003-08; Primary Completion 2007-09 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Diagnosis using KSADS | baseline, 120, 240 and 365 day follow-up.

SECONDARY OUTCOMES:
Symptomology frequency as evidenced by diary data; | daily during treatment; 3 weeks on follow-up at 240 & 365 day post randomization
Anxiety specific measure (MASC- self-report); | baseline, 120, 240 and 365 day follow-up
Disability Measure; | weekly during treatment; baseline, 120, 240 and 365 day follow-up
Child Health Questionnaire | baseline, 120, 240 and 365 day follow-up
Economic Outcome assessment | baseline, 120, 240 and 365 day follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J McGrath, PhD., Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Lingely-Pottie P, McGrath PJ. A therapeutic alliance can exist without face-to-face contact. J Telemed Telecare. 2006;12(8):396-9. doi: 10.1258/135763306779378690. PMID 17227604
- [Background] Lingley-Pottie P, McGrath PJ. Telehealth: a child and family-friendly approach to mental health-care reform. J Telemed Telecare. 2008;14(5):225-6. doi: 10.1258/jtt.2008.008001. PMID 18632994
- [Background] Lingley-Pottie P, McGrath PJ. Distance therapeutic alliance: the participant's experience. ANS Adv Nurs Sci. 2007 Oct-Dec;30(4):353-66. doi: 10.1097/01.ANS.0000300184.94595.25. PMID 18025870
- [Background] McGrath PJ, Lingley-Pottie P, Emberly DJ, Thurston C, McLean C. Integrated knowledge translation in mental health: family help as an example. J Can Acad Child Adolesc Psychiatry. 2009 Feb;18(1):30-7. PMID 19270846
- [Result] Lingley-Pottie P, McGrath PJ. A paediatric therapeutic alliance occurs with distance intervention. J Telemed Telecare. 2008;14(5):236-40. doi: 10.1258/jtt.2008.080101. PMID 18632997
- [Result] Lingley-Pottie P, Janz T, McGrath PJ, Cunningham C, MacLean C. Outcome progress letter types: parent and physician preferences for letters from pediatric mental health services. Can Fam Physician. 2011 Dec;57(12):e473-81. PMID 22170209
- [Result] McGrath PJ, Lingley-Pottie P, Thurston C, MacLean C, Cunningham C, Waschbusch DA, Watters C, Stewart S, Bagnell A, Santor D, Chaplin W. Telephone-based mental health interventions for child disruptive behavior or anxiety disorders: randomized trials and overall analysis. J Am Acad Child Adolesc Psychiatry. 2011 Nov;50(11):1162-72. doi: 10.1016/j.jaac.2011.07.013. Epub 2011 Sep 3. PMID 22024004
- See also: Family Help Program — http://www.bringinghealthhome.com/